CLINICAL TRIAL: NCT00136786
Title: Effect of Memantine Versus Bupropion on Smoking Relapse in Nicotine-Dependent Individuals
Brief Title: Effect of Memantine Versus Bupropion on Smoking Relapse in Nicotine-Dependent Individuals - 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #4725(A); R01DA017572 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco use
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Intervention 1 (Placebo Comparator): Each participant receives three consecutive interventions.
  1. Placebo
  2. Bupropion
  3. Memantine
  Interventions: Drug: Memantine
- Intervention 2 (Placebo Comparator): 1. Bupropion
  2. Memantine
  3. Placebo
  Interventions: Drug: Memantine
- Intervention 3 (Placebo Comparator): 1. Memantine
  2. Placebo
  3. Bupropion
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine

SUMMARY:
One of nicotine's effects on the body is at the level of the NMDA receptors in the brain. Memantine is a drug that also affects NMDA receptors, making it a candidate for the treatment of nicotine addiction. The purpose of this study is to evaluate the effectiveness of memantine using a laboratory model of smoking relapse in nicotine dependent volunteers. Investigators will compare the effects of memantine with bupropion, medication currently used to facilitate smoking cessation.

DETAILED DESCRIPTION:
Tobacco use is the leading preventable cause of death in the United States. Recent research on the effects of nicotine on the brain and behavior presents an opportunity to advance medication development. Neurotransmission at NMDA receptors in the brain is associated with learning and memory and has been linked to many of nicotine's effects on humans. It is possible that altering NMDA neurotransmission may be helpful in treating nicotine addiction. The goal of this study is to evaluate the effects of memantine, an NMDA receptor antagonist, using the laboratory model of smoking relapse in nicotine dependent volunteers. The effects of memantine used in combination with bupropion, a medication currently used to facilitate smoking cessation, will be compared to a placebo.

This double-blind study will consist of three phases (placebo, bupropion, and memantine). Each phase will include 10 days of outpatient medication maintenance, followed by 5 days of inpatient testing. During the outpatient phase, study visits will occur every 2 to 3 days. During the first portion of inpatient stay, participants will not be permitted to smoke. During the second portion of inpatient stay, smoking reinstatement will be modeled, as participant will have opportunity to smoke. A variety of behavioral, subjective, physiological, and performance measures will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of nicotine dependence with psychological dependence
* Smokes at least 15 cigarettes per day for the three months prior to enrollment
* Currently not seeking treatment for nicotine dependence
* Medically healthy on the basis of physical examination and medical history, vital signs, EKG, and laboratory tests
* Females must use an effective method of contraception for the duration of the study

Exclusion Criteria:

* DSM-IV diagnosis of abuse or dependence on alcohol or drugs other than nicotine
* Current Axis I diagnosis or current treatment with psychotropic medications within the three months prior to enrollment
* History of schizophrenia or other psychotic disorders, bipolar disorder, or anxiety disorders
* Currently seeking treatment for nicotine disorders
* On parole or probation
* History of seizures or head trauma with loss of consciousness, brain contusion, or fracture
* History of significant recent violent behavior
* Blood pressure greater than 150/90
* History of eating disorders
* History of allergic reaction to any of the study medications
* Pregnant

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Use of cigarettes | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States